CLINICAL TRIAL: NCT05323747
Title: Clinical Protocol for the Prospective Evaluation of a Commercially Available Hydrogel Spacer
Brief Title: Prospective Evaluation of a Commercially Available Hydrogel Spacer
Acronym: BP-008
Status: Completed | Type: Observational
Sponsor: BioProtect (Industry)
Responsible Party: Sponsor
Other Study IDs: BP-008
Record Dates: First submitted 2022-03-17; First posted 2022-04-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
Keywords: Prostate; Prostate Cancer; Spacer; Perirectal spacer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiation with Hydrogel Spacer: Males at least 18 years of age, who will be undergoing radiation therapy with a hydrogel spacer in place.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Assessment of rectal dosimetry change from pre-insertion to post-insertion in subjects with prostate cancer who have undergone radiotherapy with a hydrogel spacer.

SUMMARY:
Dosimetry efficacy evaluation of the hydrogel spacer

DETAILED DESCRIPTION:
Single arm study for evaluation of dosimetry following use of a commercially available hydrogel spacer implanted in 20 males undergoing radiotherapy to treat prostate cancer. Study will utilize pre and post gel insertion CT images to determine the endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Males
* At lease 18 years of age
* Undergoing external beam or brachy radiation therapy with a hydrogel spacer

Exclusion Criteria:

* Invasive adenocarcinoma that is extracapsular and demonstrates posterior extension

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Study Population: Prostate Cancer
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Dosimetry changes | 1 month
  Assessment of rectal radiation exposure as compared between rectal dose volume histograms calculated for pre and post Hydrogel Injection

SECONDARY OUTCOMES:
Prostate to rectum spacing | 1 month
  Prostate to rectum spacing measurement for evaluation of the perirectal distance post-hydrogel insertion

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Western Radiation Oncology, Campbell, California
  - Northern Nevada Radiation Oncology, Reno, Nevada

IPD SHARING:
Plan to Share IPD: No